CLINICAL TRIAL: NCT00318500
Title: A Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Safety and Efficacy of 75 mg and 150 mg Doses of ERB-041 on the Reduction of Symptoms Associated With Endometriosis During Treatment and Post Treatment in Reproductive-Aged Women
Brief Title: Study Evaluating the Safety and Efficacy of ERB-041 on Reduction of Symptoms Associated With Endometriosis in Reproductive-Aged Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3142A2-203
Record Dates: First submitted 2006-04-24; First posted 2006-04-26 (Estimated); Last update posted 2007-12-10 (Estimated); Status verified 2007-12

CONDITIONS: Dysmenorrhea; Dyspareunia; Endometriosis; Pelvic Pain
Keywords: Endometriosis; Dysmenorrhea; Pelvic pain; Dyspareunia
MeSH Terms: conditions — Dysmenorrhea; Dyspareunia; Endometriosis; Pelvic Pain | interventions — ERB 041

INTERVENTIONS:
Drug: ERB-041

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of two doses of ERB-041 (75 mg and 150 mg) relative to placebo on the relief of endometriosis-related symptoms (dysmenorrhea, pelvic pain, and deep dyspareunia) in reproductive aged women.

ELIGIBILITY:
Inclusion Criteria:

* Surgical diagnosis of endometriosis within the last 10 years
* Sexually active, nonpregnant, nonlactating women (18-45 years) with regular menstrual cycles who are willing to use non-hormonal contraception

Exclusion Criteria:

* Conditions requiring the use of chronic pain therapy
* Prophylactic use of analgesics to avoid endometriosis-related pain

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150
Dates: Start 2006-05; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
severity scores for dysmenorrhea, pelvic pain and deep dyspareunia from baseline through 12 weeks of treatment using the B & B scale administered by the investigator

SECONDARY OUTCOMES:
change in severity scores for pelvic tenderness and pelvic induration during 12 weeks of treatment
change in rescue medication use
change in health related quality of life questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For United Kingdom, ukmedinfo@wyeth.com; Trial Manager, Principal Investigator — For Australia and Hong Kong, medinfo@wyeth.com; Trial Manager, Principal Investigator — For South Africa, ZAFinfo@wyeth.com; Trial Manager, Principal Investigator — For Belgium, trials-BEL@wyeth.com; Trial Manager, Principal Investigator — For Canada, clintrialparticipation@wyeth.com
Locations (65):
- United States (44):
  - Montgomery, Alabama
  - Chandler, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - San Francisco, California
  - Vista, California
  - Denver, Colorado
  - New Britain, Connecticut
  - Clearwater, Florida
  - New Port Richey, Florida
  - Plantation, Florida
  - Venice, Florida
  - West Palm Beach, Florida
  - Marietta, Georgia
  - Idaho Falls, Idaho
  - Oak Brook, Illinois
  - Evansville, Indiana
  - Reno, Nevada
  - Lawrenceville, New Jersey
  - Durham, North Carolina
  - New Bern, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Miamisburg, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Abington, Pennsylvania
  - Lansdale, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Columbia, South Carolina
  - Greenville, South Carolina
  - Bristol, Tennessee
  - Chattanooga, Tennessee
  - Memphis, Tennessee
  - Corpus Christi, Texas
  - San Antonio, Texas
  - West Valley City, Utah
  - Norfolk, Virginia
  - Richmond, Virginia
  - Virginia Beach, Virginia
  - Renton, Washington
  - Madison, Wisconsin
- Australia (4):
  - Randwick, New South Wales
  - Sydney, New South Wales
  - Richmond, Victoria
  - Nedlands, Western Australia
- Herestraat, Leuven, Belgium
- Canada (7):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Halifax, Nova Scotia
  - London, Ontario
  - Toronto, Ontario
  - Saskatoon, Saskatchewan
- Hong Kong, Hong Kong
- South Africa (4):
  - Cape Town, Capetown
  - Port Elizabeth, Eastern Cape
  - Roodepoort, Jgb Gauteng
  - Durban, KwaZulu-Natal
- United Kingdom (4):
  - Nottingham, Nottinghamshire
  - Glasgow, Scotland
  - Sheffield, South Yorshire
  - Swindon, Wiltshire